CLINICAL TRIAL: NCT00609063
Title: The Effect of Statins on Skeletal Muscle Function
Brief Title: The Effect of Statin Medications on Muscle Performance (The STOMP Study)
Acronym: STOMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 552; R01HL081893-01A2 (NIH); 1R01HL081893-01A2 (NIH); 105-0342
Record Dates: First submitted 2008-01-25; First posted 2008-02-06 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: Hydroxymethylglutaryl-CoA Reductase Inhibitors; Muscular Diseases
Keywords: Statins; Myalgia; Muscle Cramp
MeSH Terms: conditions — Muscular Diseases; Myalgia; Muscle Cramp | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive atorvastatin for 6 months.
  Interventions: Drug: Atorvastatin
- 2 (Placebo Comparator): Participants will receive matching placebo for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — 80-mg atorvastatin capsules taken daily for 6 months
  Other Names: Lipitor
  Arms: 1
Drug: Placebo — Placebo capsules taken daily for 6 months
  Arms: 2

SUMMARY:
Statins are a group of medications that are used to lower cholesterol levels. Although serious side effects are rare, some people taking statins experience muscle pain or weakness. This study will evaluate the number of people who experience mild muscle complaints and will determine the effect of statins on skeletal muscle strength, endurance, and aerobic exercise performance.

DETAILED DESCRIPTION:
Statins are the most effective medications for reducing high cholesterol levels. They are extremely well tolerated by the majority of people but can produce a variety of muscle-related side effects in some people. Of these side effects, the most serious is rhabdomyolysis, which involves muscle fiber damage that can begin as muscle pain and progress to a loss of muscle cells, kidney failure, and death. While rhabdomyolysis is extremely rare, some people experience the more common muscle-related side effects of statins, such as muscle pain (known as "myalgia"), cramps, and weakness. These more common side effects warrant attention because they may limit the use of statins, affect mobility, and increase the risk of injury in older individuals. Also, the term "muscle weakness," often used by patients and their doctors, is not well defined and can refer to a wide range of complaints from simple fatigue to an actual inability to perform activities of daily living. It is important to describe and quantify in more detail the muscle-related side effects associated with statins. The purpose of this study is to determine the incidence of statin-induced mild muscle complaints and to determine the effect of statins on skeletal muscle strength, endurance, and aerobic exercise performance.

This study will enroll healthy people who have never received statin medications. First, participants will attend three study visits over a period of 2 weeks. These study visits will include blood collection, questionnaires on physical activity and pain, vital sign measurements, and body measurements, including height, weight, and head circumference. Participants will also complete two cardiopulmonary exercise stress tests on a treadmill and will undergo arm and leg strength testing. Some participants may undergo a muscle biopsy. Participants will then be randomly assigned to receive either 80 mg of atorvastatin or placebo on a daily basis for 6 months. Blood will be collected again at Month 3. At Month 6, participants will attend two study visits for repeat baseline measurements. All participants will be contacted by phone every other week during the 6-month treatment period to monitor adverse events and medication compliance.

ELIGIBILITY:
Inclusion Criteria:

* Statin-naive (i.e., has never taken statins before)

Exclusion Criteria:

* Previous use of statins
* Current treatment with cholesterol- or triglyceride-lowering drugs
* Impaired liver or kidney function
* Untreated hypothyroidism or hyperthyroidism
* Treatment with other medications known to increase risk of myopathy in atorvastatin-treated patients (e.g., cyclosporine, azithromycin, erythromycin, azole antifungals, fusidic acid)
* Existing infection requiring treatment with antibiotic therapy
* Consumption of greater that 1 quart of grapefruit juice per day
* Documented history of neuroleptic malignant syndrome
* Inherited muscle disorders or myopathy
* Known sickle cell trait
* Cancer within the 5 years prior to study entry
* Diabetes
* Currently being treated for high blood pressure
* Coronary artery disease
* Peripheral vascular disease
* Physical disability or previous injury that prevents safe exercise testing
* Pregnant or breastfeeding

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2008-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Myopathy frequency | Measured every other week
Arm isokinetic force at 60 degrees per second | Measured at Month 6
Leg isokinetic force at 60 degrees per second | Measured at Month 6
Handgrip isometric force | Measured at Month 6
Leg dynamic endurance | Measured at Month 6
Maximal aerobic power | Measured at Month 6

SECONDARY OUTCOMES:
Structural differences in the muscle samples obtained from symptomatic and asymptomatic participants | Measured after 2 weeks of symptom persistence
Skeletal muscle gene expression in muscle samples obtained from symptomatic and asymptomatic participants | Measured after 2 weeks of symptom persistence

CONTACTS AND LOCATIONS:
Overall Officials: Paul D. Thompson, MD, Principal Investigator — Hartford Hospital
Locations (3):
- United States (3):
  - Hartford Hospital, Hartford, Connecticut
  - University of Connecticut, Storrs, Connecticut
  - University of Massachusetts, Amherst, Massachusetts

REFERENCES:
- [Derived] Taylor BA, Dager AD, Panza GA, Zaleski AL, Meda S, Book G, Stevens MC, Tartar S, White CM, Polk DM, Pearlson GD, Thompson PD. The effect of high-dose atorvastatin on neural activity and cognitive function. Am Heart J. 2018 Mar;197:166-174. doi: 10.1016/j.ahj.2017.10.027. Epub 2017 Dec 6. PMID 29447778
- [Derived] Ballard KD, Taylor BA, Capizzi JA, Grimaldi AS, White CM, Thompson PD. Atorvastatin Treatment Does Not Alter Pulse Wave Velocity in Healthy Adults. Int Sch Res Notices. 2014 Nov 13;2014:239575. doi: 10.1155/2014/239575. eCollection 2014. PMID 27351006
- [Derived] Ballard KD, Parker BA, Capizzi JA, Grimaldi AS, Clarkson PM, Cole SM, Keadle J, Chipkin S, Pescatello LS, Simpson K, White CM, Thompson PD. Increases in creatine kinase with atorvastatin treatment are not associated with decreases in muscular performance. Atherosclerosis. 2013 Sep;230(1):121-4. doi: 10.1016/j.atherosclerosis.2013.07.001. Epub 2013 Jul 13. PMID 23958263
- [Derived] Parker BA, Capizzi JA, Grimaldi AS, Clarkson PM, Cole SM, Keadle J, Chipkin S, Pescatello LS, Simpson K, White CM, Thompson PD. Effect of statins on skeletal muscle function. Circulation. 2013 Jan 1;127(1):96-103. doi: 10.1161/CIRCULATIONAHA.112.136101. Epub 2012 Nov 26. PMID 23183941
- [Derived] Parker BA, Capizzi JA, Augeri AL, Grimaldi AS, Michael White C, Thompson PD. Atorvastatin increases exercise leg blood flow in healthy adults. Atherosclerosis. 2011 Dec;219(2):768-73. doi: 10.1016/j.atherosclerosis.2011.09.049. Epub 2011 Oct 4. PMID 22018642